CLINICAL TRIAL: NCT02560467
Title: Perfusion Imaging With Myocardial Contrast Echocardiography in HCM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jonathan R. Lindner, MD, Professor, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15158
Record Dates: First submitted 2015-09-22; First posted 2015-09-25 (Estimated); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — Caves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with HCM (Experimental): This is a prospective, non-blinded single center study. Subjects with known HCM with variant will be recruited. MCE at rest and during vasodilator stress will be performed. Full echocardiography including for diastolic function and regional strain imaging will also be performed. Patient history and questionnaires will be used for evaluation of symptoms and arrhythmias.
  Interventions: Drug: Echo and myocardial contrast echocardiography perfusion imaging

INTERVENTIONS:
Drug: Echo and myocardial contrast echocardiography perfusion imaging — Myocardial blood flow will be assessed by myocardial contrast echo. Perfusion at rest and stress will be quantified and compared to patient sx, degree of dysfunction on echo strain imaging, and degree of fibrosis on magnetic resonance imaging (when available) that was ordered as part of routine clinical care.
  Myocardial contrast echocardiography will be performed by intravenous administration of ultrasound contrast agent (Definity or Lumason) using FDA-approved dose limits. Vasodilator stress during MCE imaging will be performed using regadenoson at FDA-approved doses.

SUMMARY:
The objective of this study is to determine whether myocardial contrast echocardiography in patients with cardiomyopathy (HCM) can detect resting hypo-perfusion due to fibrosis or stress induced perfusion defects due to associated abnormalities in intramyocardial arteries and the microcirculation. A secondary aim will be to determine whether abnormalities in perfusion are associated with either severity of symptoms (chest pain and dyspnea), presence of arrhythmias, and regional function of the septum.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Established diagnosis of HCM

Exclusion Criteria:

* Known history of coronary or peripheral artery disease
* History of myocardial infarction
* Pregnant or lactating females
* Hypersensitivity to any ultrasound contrast agent
* Evidence right-to-left or bi-directional intracardiac shunt
* Moderate or greater valve disease other than from HCM (systolic anterior motion of the mitral valve)
* History of septal ablation or myectomy
* Hemodynamic instability
* Pacemaker dependent heart rhythm

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-09-15 (Estimated)

PRIMARY OUTCOMES:
Myocardial perfusion (ml/min/g) in the hypertrophied segment on myocardial contrast echo | One hour
  Myocardial contrast echo will be used to measure myocardial perfusion in ml/min/g of tissue in the hypertrophied segment. The data will be analyzed both in terms of absolute value of ml/min/g and also as a ration to normal tissue.
Myocardial blood flow reserve in the hypertrophied segment on myocardial contrast echo | One hour
  Myocardial blood flow reserve on myocardial contrast echo (ratio of flow during hyperemia to rest) will be calculated for the hypertrophied segment and expressed as an absolute value and relative to normal segments.

SECONDARY OUTCOMES:
Spatial distribution of blood flow on myocardial contrast echocardiography | One hour
  Myocardial contrast echocardiography performed at baseline will be analyzed using mathematical algorithms that define how "homogenous" or "heterogenous" blood flow distribution is in the hypertrophied segment. These values will be described by wavelet energy levels (dimensionless).

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Derived] Roldan P, Ravi S, Hodovan J, Belcik JT, Heitner SB, Masri A, Lindner JR. Myocardial contrast echocardiography assessment of perfusion abnormalities in hypertrophic cardiomyopathy. Cardiovasc Ultrasound. 2022 Sep 19;20(1):23. doi: 10.1186/s12947-022-00293-2. PMID 36117179